CLINICAL TRIAL: NCT00786383
Title: Phase 1 Study of Every Other Week Anti-Vascular Endothelial Growth Factor Receptor 2 (VEGFR-2) Monoclonal Antibody IMC-1121B in Patients With Advanced Solid Tumors Who Have Not Responded To Standard Therapy
Brief Title: Study of IMC-1121B in Patients With Advanced Solid Tumors Not Responding To Standard Therapy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13919; CP12-0402 (Other: ImClone Systems); I4T-IE-JVBN (Other: Eli Lilly and Company)
Record Dates: First submitted 2008-11-04; First posted 2008-11-06 (Estimated); Last update posted 2013-08-19 (Estimated); Status verified 2013-08

CONDITIONS: Cancer
Keywords: Phase I; cancer; solid tumors; 1121B; VEGFR-2; Anti-Vascular Endothelial Growth Factor Receptor 2
MeSH Terms: conditions — Neoplasms | interventions — Ramucirumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- IMC-1121B (Experimental): IMC-1121B injectable solution at a concentration of 5 mg/mL in single-use vials containing 100 mg/20 mL or 250 mg/50 mL of product, administered intravenously at an initial dose of 6 mg/kg.A minimum of three patients will be enrolled into each cohort. When all patients complete a cohort, dose escalation to the next cohort will occur.
  Interventions: Biological: IMC-1121B; Biological: 1121B

INTERVENTIONS:
Biological: IMC-1121B — Cohort 1
  6 mg/kg I.V., once every other week for 4 weeks
Biological: 1121B — Cohort 2
  8mg/kg I.V., once every other week for 4 weeks
Biological: 1121B — Cohort 3
  10 mg/kg I.V., once every other week for 4 weeks
Biological: 1121B — Cohort 4
  15 mg/kg I.V., once every 3 weeks for 6 weeks
Biological: 1121B — Cohort 5
  20 mg/kg I.V., once every 3 weeks for 6 weeks

SUMMARY:
We are conducting a research study for tumors that have not responded to prior treatment. The subject will receive an investigational drug called IMC-1121B. ImClone LLC, the maker of IMC-1121B, is running this research study.

We believe that IMC-1121B blocks the growth factors made by the cancer cells, so new blood vessels do not grow. It is believed that without the new blood vessels, the cancer or tumor will not get the oxygen and food that it needs to grow. This may stop the cancer from growing or spreading and the tumor cells may die. Since normal blood vessels have already formed in adults, it might be possible to stop tumor growth without harming normal cells.

DETAILED DESCRIPTION:
We are conducting a research study for tumors that have not responded to prior treatment. The subject will receive an investigational drug called IMC-1121B. ImClone LLC, the maker of IMC-1121B, is running this research study.

In order for a cancer to grow, it needs blood vessels to bring to it oxygen and food. Cancer cells can make growth factors that cause the abnormal growth of new blood vessels. This is called angiogenesis. Normally, new blood vessels do not grow in adults. Angiogenesis inhibitors are drugs that may prevent abnormal growth of blood vessels to tumors. IMC-1121B is an angiogenesis inhibitor. We believe that IMC-1121B blocks the growth factors made by the cancer cells, so new blood vessels do not grow. It is believed that without the new blood vessels, the cancer or tumor will not get the oxygen and food that it needs to grow. This may stop the cancer from growing or spreading and the tumor cells may die. Since normal blood vessels have already formed in adults, it might be possible to stop tumor growth without harming normal cells.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histopathologically-documented, measurable or evaluable (non-measurable), advanced primary or recurrent solid tumors who have not responded to standard therapy or for whom no standard therapy is available
* Eastern Cooperative Oncology Group (ECOG) performance status score of ≤2 at study entry.
* Able to provide written informed consent.
* A life expectancy of >3 months.
* Adequate hematologic function, as defined by:

  * an absolute neutrophil count ≥1500/mm3
  * a hemoglobin level ≥10 gm/dL
  * a platelet count ≥100,000/mm3
* Adequate hepatic function, as defined by:

  * a total bilirubin level ≤1.5 x the upper limit of normal (ULN)
  * aspartate transaminase (AST) and alanine transaminase (ALT) levels ≤2.5 x the ULN or ≤5 x the ULN if known liver metastases
* Adequate renal function, as defined by a serum creatinine level ≤1.5 x the ULN.
* Use of effective contraception , if procreative potential exists.
* Adequate recovery from recent surgery, chemotherapy, and radiation therapy. At least 28 days must have elapsed from major surgery, prior chemotherapy, prior treatment with an investigational agent or device, or prior radiation therapy
* Accessible for treatment and follow-up. Patients enrolled in this trial must be treated at the participating center.

Exclusion Criteria:

* Patients with large centrally-located pulmonary lesions adjacent to or invading large blood vessels.
* Patients who have had chemotherapy or therapeutic radiotherapy within 28 days (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or patients with ongoing side effects ≥ grade 2 due to agents administered more than 28 days earlier.
* Prior left chest wall radiotherapy or a cumulative anthracycline dose ≥300 mg/m2 (if the ejection fraction is within normal institutional limits, the patient can be enrolled).
* Any concurrent malignancy other than non-melanomatous skin cancer or carcinoma in situ of the cervix. Patients with a previous malignancy but without evidence of disease for ≥3 years will be allowed to enter the trial.
* Uncontrolled intercurrent illness including, but not limited to:

  * ongoing or active infection requiring parenteral antibiotics
  * symptomatic congestive heart failure (class III or IV of the New York Heart Association classification for heart disease)
  * unstable angina pectoris, angioplasty, stenting, or myocardial infarction within 6 months
  * uncontrolled hypertension (systolic blood pressure ≥160 mm Hg, diastolic blood pressure >100 mm Hg, found on two consecutive measurements separated by a 1-week period despite adequate medical support)
  * clinically significant cardiac arrhythmia (multifocal premature ventricular contractions, bigeminy, trigeminy, ventricular tachycardia that is symptomatic or requires treatment or asymptomatic sustained ventricular tachycardia)
  * uncontrolled diabetes
  * psychiatric illness/social situations that would compromise patient safety or limit compliance with study requirements
  * patients with symptomatic brain metastases (patients with a history of brain metastases must have received definitive surgery or radiotherapy, be clinically stable, and not taking steroids; anticonvulsants are allowed)
* A serious or nonhealing active wound, ulcer, or bone fracture.
* Known human immunodeficiency-positivity.
* A major surgical procedure, an open biopsy, or a significant traumatic injury within 28 days prior to treatment.
* Current or recent use (within 28 days) of a thrombolytic agent.
* Current or recent use (within 28 days) of full-dose warfarin (an exception is low-dose warfarin to maintain patency of preexisting, permanent, indwelling intravenous (i.v.) catheters; for patients receiving warfarin, the international normalized ratio [INR] should be <1.5). Patients requiring heparin are excluded.
* Chronic daily treatment with aspirin (>325 mg/day) or nonsteroidal anti-inflammatory medications known to inhibit platelet function (cyclooxygenase-2 [COX-2] inhibitors are permitted).
* A history or clinical evidence of a deep venous or arterial thrombosis (including pulmonary embolism) within the last 6 months prior to study entry.
* Proteinuria ≥1+ by routine urinalysis (patients with a protein value of ≤500 mg confirmed by a 24-hour urine collection are eligible).
* Pregnant (confirmed by serum beta human chorionic gonadotropin [βHCG]) or breast feeding.
* Prior treatment with bevacizumab or other agents specifically targeting VEGF ligand or receptor within 6 weeks of study entry.
* Monoclonal antibodies within 6 weeks of study entry.
* Positive anti-IMC-1121B antibody response.
* A history of allergic reactions to monoclonal antibodies or other therapeutic proteins.
* The subject is the investigator, sub-investigator, or anyone directly involved in the conduct of the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2006-02; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Number of participants with Adverse Events (AEs) | 8 Weeks
Maximum Tolerated Dose | 8 Weeks

SECONDARY OUTCOMES:
Maximum concentration (Cmax), cohorts 1, 2, 3, 4, and 5 | 8 Weeks
Minimum concentration (Cmin), cohorts 1, 2, 3, 4, and 5 | 8 Weeks
Area under concentration (AUC), cohorts 1, 2, 3, 4, and 5 | 8 Weeks
Half-life (t 1/2), cohorts 1, 2, 3, 4, and 5 | 8 Weeks
Clearance (Cl) rate drug is completely removed, cohorts 1, 2, 3, 4, and 5 | 8 Weeks
Volume of distribution (Vss) at steady state, cohorts 1, 2, 3, 4, and 5 | 8 Weeks
Serum Anti-IMC-1121B Antibody Assessment (immunogenicity) | 8 Weeks
Change in tumor size from Baseline Measurement | 8 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Chair — Eli Lilly and Company
Locations (3):
- United States (3):
  - ImClone Investigational Site, Indianapolis, Indiana
  - ImClone Investigational Site, Durham, North Carolina
  - ImClone Investigational Site, Philadelphia, Pennsylvania

REFERENCES:
- [Derived] Chiorean EG, Hurwitz HI, Cohen RB, Schwartz JD, Dalal RP, Fox FE, Gao L, Sweeney CJ. Phase I study of every 2- or 3-week dosing of ramucirumab, a human immunoglobulin G1 monoclonal antibody targeting the vascular endothelial growth factor receptor-2 in patients with advanced solid tumors. Ann Oncol. 2015 Jun;26(6):1230-1237. doi: 10.1093/annonc/mdv144. Epub 2015 Mar 18. PMID 25787923